CLINICAL TRIAL: NCT05032131
Title: Cell Therapy for Inclusion Body Myositis (IBM) by Muscle Injection of Autologous Uncultured Adipose-Derived Stromal Vascular Fraction (ADSVF): a Phase I Trial
Brief Title: Cell Therapy for IBM by Muscle Injection of ADSVF
Acronym: ADSVF-in-IBM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP180593; 2020-005876-36 (EudraCT Number)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Inclusion Body Myositis
Keywords: Inclusion Body Myositis; Cell Therapy; ADSVF
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Group 1:
  Patients treated by sirolimus since at least 6 months (but still disabled)
  Group 2:
  Patients currently (for at least 3 months) without specific treatment for inclusion myositis
  Interventions: Biological: ADSVF

INTERVENTIONS:
Biological: ADSVF — Group 1 and 2 : Escalating dose of ADSVF injection (5 millions of cells, 10 millions of cells and 20 millions of cells).

SUMMARY:
Inclusion Body Myositis is a slowly but disabling myopathy, the most frequent in patients over 50 years old. No treatments (in particular immunosuppressive) are known to be efficient.

Autologous uncultured adipose-derived stromal vascular fraction (ADSVF) is recognized as an easily accessible (by a standard liposuction to obtain adipose tissue, from which ADSVF are isolated by centrifugation), safe and well tolerated source of cells with angiogenic, anti-inflammatory, immunomodulatory and regenerative properties. The purpose of our ADSVF in IBM phase I trial is to evaluate, for the first time in human diseased muscle, first the tolerance of autologous ADSVF cells locally injected in affected forearm muscles and second their capability to repair those muscles. With always the goals of tolerance first and second muscle repair, we will recruit in parallel two groups of IBM patients: the first treated by sirolimus since at least 6 months (but still disabled) and the second currently (for at least 3 months) without specific treatment for inclusion myositis.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the tolerance of escalating doses of ADSVF, one month after intramuscular injection in the finger flexors, in the non-dominant forearm. The second objective of this study is to evaluate the efficacy in term of muscle repair (regenerative properties of ADSVF) and in term of muscle inflammation control, during 6 months, by functional strength tests, quantitative MRI and PBMC monitoring. This research is a phase I trial evaluating first the tolerance and second the efficacy of 3 escalating doses of ADSVF intramuscularly injected in the non-dominant forearm. The volume of injection will be of 1 ml in each of the 5 sites of the finger flexoses, in line at 1 cm apart, for a total dose of 5 millions (low dose) or 10 millions (intermediate dose) or 20 millions (high dose) of viable nucleated cells.These doses are chosen because of the perfect tolerance of intra-muscle injection of (in average) one million ADSVF per millilitre, with a total dose of viable nucleated cells injected between 2.5 and 8.6 millions.The cell treatment will be prepared from autologous uncultured Adipose-Derived Stromal Vascular Fraction (ADSVF) isolated by centrifugation of adipose tissue obtain by liposuction. The study population will be adult patients suffering of an Inclusion Body Myositis (IBM) fulfilling the Lloyd criteria treated by sirolimus since at least 6 months (but still disabled) - who are part of group 1 or currently (for at least 3 months) without specific treatment for inclusion myositis - who are part of group 2. The main inclusion criteria are : Patients: with an age ≥ 45 and ≤ 80 years old, with IBM defined by the Lloyd criteria: muscle weakness of finger flexors or quadriceps, and endomysial inflammatory infiltrates on muscle biopsy, and presence of invaded fibers or rimmed vacuoles on muscle biopsy, who gave their written informed consent, affiliated to a social security regime (expected AME) ; and for: group 1: treated by sirolimus since at least 6 months (but still disabled ) - group 2: currently (for at least 3 months) without specific treatment for inclusion myositis - group 2. The duration of participation of the patients will be 7 months, included one month between maximum the inclusion visit and the injection visit, and 6 month of follow-up periof after ADSVF injection.

ELIGIBILITY:
Inclusion Criteria:

* With an age ≥ 45 and ≤ 80 yo.
* Man or menopausal woman. - With IBM defined by the Lloyd criteria (Lloyd et al., 2014): muscle weakness of finger flexors or quadriceps, and endomysial inflammatory infiltrates on muscle biopsy, and presence of invaded fibers or rimmed vacuoles on muscle biopsy.
* Who gave their written informed consent
* Affiliated to a social security regime (expected AME) And for: -group 1: treated by sirolimus since at least 6 months (but still disabled ) - group 2: currently (for at least 3 months) without specific treatment for inclusion myositis.

Exclusion Criteria:

* Impossibility to walk 10 meters
* Grip evaluated by MRC5 MMT at 0 OR 1.
* Body mass index < 18
* Not able to stop any anticoagulant, or antiaggregant drugs within the week before and the 48 hours before the liposuction
* Severe respiratory insufficiency (FVC < 50% and/or FEV1 < 50%)
* Severe chronic kidney disease (Estimated Glomerular Filtration Rate < 15 ml/min and/or proteinuria > 0.5 g/24h)
* Cancer non in remission (necessitating specific treatment) during the past 12 months
* Connective Tissue Disease non in remission (necessitating specific treatment) during the past 12 months - Bone marrow transplantation
* Connective Tissue disease non in remission (necessitating specific treatment) during the past 12months - Immunosuppressive drugs except sirolimus, ongoing or stopped in less than 3 months
* Polyvalent immunoglobulins (IV or sub-cut) ongoing or stopped in less than 3 months
* Any biotherapies (mAbs) such as ant-CD20, CTLA4Ig, anti-TNF, anti-IL6R, anti-IL1 etc… ongoing or stopped in less than 6 months.
* Seropositivity for HIV, HCV or HBV
* Contraindication to muscle MRI
* Contraindications to the liposuction: eg coagulation disorders, etc… - Contraindications to anaesthetics
* Documented conventional antibiotics severe allergy such as ß-lactam (cephalosporin), cyclins, macrolides (for example metronidazole), quinolones
* Participation in another trial (Jardé 1 or Jardé 2)
* Legal protection (curatorship or tutorship) or safety measure

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
In each group, tolerance of escalating doses (3+3) of ADSVF in the non-dominant forearm | Days 0 (day of the injection) to day 30
  By determining the dose-limiting toxicity (DLT)

SECONDARY OUTCOMES:
In each group, tolerance of escalating doses (3+3) of ADSVF in the non-dominant forearm | Days 0 (day of the injection) to 6 months (end of participation)
  By research of adverse events
In each group, efficacy in term of muscle repair (regenerative properties of ADSVF) | At day 30, 3 month and 6 month
  Functional muscle evaluations
In each group, efficacy in term of muscle repair (regenerative properties of ADSVF) | At 6 month
  Muscle mass, fatty replacement and inflammation by quantitative NMRI
In each group, evaluation of muscle inflammation control | At 6 month
  Immunomonitoring of the peripheral blood mononuclear cells (PBMC)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Benveniste, Professor, Principal Investigator — APHP
Locations (1):
- Olivier BENVENISTE, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal